CLINICAL TRIAL: NCT01815567
Title: The Effects of Blood Pressure on Cognitive Function: Examining the Use of Bedside Neuropsychological Testing During Acute Hypertensive Events
Brief Title: DETECT and Retinal Outcomes in Hypertension
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Tamara Espinoza, MD, Assistant Professor, Emory University
Other Study IDs: IRB00060043
Record Dates: First submitted 2012-09-20; First posted 2013-03-21 (Estimated); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Hypertension; Retinal Disorder; Cognitive Impairment
Keywords: Hypertension; Retinal Disorder; Cognitive impairment
MeSH Terms: conditions — Hypertension; Retinal Diseases; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- controlled hypertension: hypertension with medication controlled
- uncontrolled hypertension: non-controlled hypertension
- hypertensive urgency: hypertensive urgency no previous history or antihypertensives
- asymptomatic normotensive: asymptomatic normotensive control group

SUMMARY:
The purpose of this study is to study the impact of blood pressure on cognitive performance.

DETAILED DESCRIPTION:
Four groups will be evaluated for possible impact of blood pressure on cognitive performance and retinal damage.

ELIGIBILITY:
Inclusion Criteria:

1. Patients triaged to the Grady Memorial Hospital Emergency Department or Marcus Trauma Unit
2. Age >18 and <65
3. Documented history of hypertension plus one or more of the following:

   * current antihypertensive use with controlled blood pressure
   * elevated Emergency Department systolic blood pressure or diastolic blood pressure
   * OR -
4. Acutely elevated Emergency Department systolic blood pressure or diastolic blood pressure on 2 separate Emergency Department measurements in the absence of a history of hypertension

   * OR -
5. Normal systolic blood pressure or diastolic blood pressure in the absence of hypertension.

Exclusion Criteria:

1. Non-English speaking
2. Pre-visit cognitive impairment
3. Physical or psychological impairments that would prohibit comprehension and completion of DETECT testing
4. Inability to obtain adequate fundoscopic photos
5. Acute intoxication, altered mental status, or head injury within the last 6 months
6. Opiate or benzodiazepine administration by treating providers
7. Clinical condition not allowing testing.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Emergency department patients that meet the inclusion/exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 234 (Actual)
Dates: Start 2012-11; Primary Completion 2020-07-15 (Actual); Study Completion 2020-07-15 (Actual)

PRIMARY OUTCOMES:
DETECT neurocognitive outcome scores (Z-scores) in association with blood pressure measures and retinal pathology (isolated retinal hemorrhage, grade III/IV hemorrhagic retinopathy) | 12 months
  We aim to determine the correlation (if any) between the severity of blood pressure and DETECT neurocognitive outcomes as well as the correlation (if any) between known Hypertensive retinal disease and DETECT neurocognitive outcomes. Appropriate statistical analysis will be performed to compare clinical retinal findings, BP values, and DETECT neurocognitive test outcomes.
  Subject level data will only be collected on the day of Emergency Department presentation. Subjects will not be followed after their initial enrollment. The study duration is projected for 12 months

SECONDARY OUTCOMES:
Variance of DETECT scores (Z-score) attributed to reading level | One year study periord (12 months)

CONTACTS AND LOCATIONS:
Overall Officials: Tamara Espinoza, MD, Principal Investigator — Emory University
Locations (1):
- Grady Memorial Hospital, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No